CLINICAL TRIAL: NCT00617188
Title: Phase II Trial of Fulvestrant in Treatment of Recurrent Ovarian Carcinoma
Brief Title: Fulvestrant in Treating Patients With Recurrent Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582821; UMN-2007LS003 (Other: Clinical Trials Office, University of Minnesota); UMN-WCC-49 (Other: Women's Cancer Center, University of Minnesota); UMN-0612M97626 (Other: IRB, University of Minnesota); IRUSFULV0062 (Other: AstraZeneca)
Record Dates: First submitted 2008-02-14; First posted 2008-02-15 (Estimated); Results first posted 2010-03-17 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer
Keywords: recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fulvestrant (Experimental): Fulvestrant 500 milligrams (mg) Day 1; 250 mg Day 1, 29 and every 28 days thereafter.
  Interventions: Drug: Fulvestrant

INTERVENTIONS:
Drug: Fulvestrant — Fulvestrant, 500 milligrams (mg) intramuscularly (IM) on Day 1, 250 mg IM on Day 15, and 250 mg IM on Day 29 and every 28 days thereafter until either intolerance or disease progression.
  Other Names: Faslodex

SUMMARY:
RATIONALE: Estrogen can cause the growth of ovarian epithelial cancer cells. Hormone therapy using fulvestrant may fight ovarian cancer by blocking the use of estrogen by the tumor cells.

PURPOSE: This phase II trial is studying how well fulvestrant works in treating patients with recurrent ovarian epithelial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the 90-day clinical benefit (defined as the sum of complete responses, partial responses, and stable disease) in patients with recurrent ovarian epithelial cancer treated with single agent fulvestrant.

Secondary

* To establish the time to termination of treatment (due to all causes including progression and intolerance) for patients treated with this drug.
* To describe the toxicities observed in patients treated with this drug.
* To evaluate the quality of life of patients treated with this drug.
* To determine the effect that prolonged estrogen receptor antagonism has on markers of bone mineral turnover.

OUTLINE: Patients receive fulvestrant intramuscularly on days 1 and 15 of course 1 and then on day 1 of all subsequent courses. Treatment repeats every 28 days for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients in continued response at the end of 1 year may continue treatment at the discretion of the treating physician.

Urinary N-telopeptide and serum skeletal-specific alkaline phosphatase are assessed at baseline and at 1, 3, and 6 months during study to determine the influence of estrogen blockade on bone mineral turnover.

Quality of life is assessed at baseline and every 3 months during treatment, and at the end of treatment using The Functional Assessment of Cancer Therapy - Ovarian (FACT-O) cancer questionnaire.

After completion of study treatment, patients are followed at approximately 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial carcinoma

  * Recurrent or persistent disease

    * Must have received greater than or equal to (≥) 2 prior cytotoxic chemotherapy regimens, including ≥ 1 platinum-containing regimen
  * Disease not amenable to curative treatment with surgery and/or radiotherapy
* Must have measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST) and/or a serum cancer antigen 125 (CA-125) level that is rising and meets 1 of the following criteria:

  * Serum CA-125 level greater than (>) upper limit of normal (typically 35 μ/mL) on two evaluations at least 2 weeks apart
  * Serum CA-125 level less than (<) 35 μ/mL but has risen progressively > 200% over successive specimens ≥ 2 weeks apart
* Estrogen receptor-positive tumor
* Gynecologic Oncology Group (GOG) performance status 0-3
* Platelet count ≥ 50 x 10^9/Liter
* Serum creatinine less than or equal to (≤) 2.5 mg/deciliter
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) ≤ 3 times upper limit of normal (ULN)
* alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5 times ULN (≤ 5 times ULN in the presence of liver metastases)
* Alkaline phosphatase ≤ 3 times ULN
* Prothrombin time-International Normalized Ratio (INR) ≤ 1.6
* Not pregnant or nursing
* Negative pregnancy test
* Must be sterile or fertile patients must use effective contraception (i.e., double method including ≥ 1 barrier, injectable, implantable, condoms plus spermicide)
* Prior malignancy allowed provided the patient has been disease-free for ≥ 5 years

  * Patients with previously diagnosed basal cell skin cancer are eligible immediately after completing therapy
* No history of bleeding (i.e., disseminated intravascular coagulation or clotting factor deficiency)
* No documented sensitivity to active or inactive excipients of fulvestrant (i.e., castor oil or mannitol)
* Recovered from the effects of prior surgery, radiotherapy, and/or chemoradiotherapy
* At least 3 weeks since prior chemotherapy
* At least 3 weeks since prior complete radiotherapy regimen alone or chemoradiotherapy

  * An incomplete radiotherapy regimen (< 500 Gray) is allowed within the 3-week time frame

Exclusion Criteria:

* Concurrent hormone replacement therapy
* Prior long-term anticoagulation therapy other than anti-platelet therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Argenta, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Argenta PA, Thomas SG, Judson PL, Downs LS Jr, Geller MA, Carson LF, Jonson AL, Ghebre R. A phase II study of fulvestrant in the treatment of multiply-recurrent epithelial ovarian cancer. Gynecol Oncol. 2009 May;113(2):205-9. doi: 10.1016/j.ygyno.2009.01.012. Epub 2009 Feb 23. PMID 19239974

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 additional patients were enrolled, but were never treated.
Groups:
- Fulvestrant Treatment: Patients who met Inclusion Criteria and received at least 1 dose of study drug (Fulvestrant 500 mg Day 1; 250 mg Day 1, 29 and every 28 days thereafter)
Period: Overall Study
Arm/Group | Fulvestrant Treatment
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Secondary Outcome: Patients' Overall 90-Day Clinical Response as Measured by Modified Response Evaluation Criteria in Solid Tumors (Rustin)
Description: Defined by the sum of Complete Responses (CR), Partial Responses (PR) and Stable Disease (SD) in patients treated with fulvestrant. CR=normalization of serum CA-125 level from 2 initially elevated samples, PR=>or=50% decrease in serum CA-125 level from 2 initially elevated samples, Progressive Disease (PD)=CA-125 two times the upper limit of normal on 2 occasions (if previously normalized) OR CA-125 two times nadir (lowest value) on 2 occasions if elevated at initiation of treatment, SD=not CR, PR or PD.
Time Frame: Day 90
Measure: Number; unit: Participants
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Participants
  Stable Disease | 13
  Progressive Disease (>= 20% increase/new lesions) | 13

2. Secondary Outcome: Median Number of Days to Treatment Termination
Description: Time is determined from first dose to termination due to all causes.
Time Frame: Up to 373 Days
Measure: Median (Full Range); unit: Days
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Days | 62 [5 to 373]

3. Secondary Outcome: Mean Scores - Quality of Life Assessment
Description: Functional Assessment of Cancer Therapy-Ovarian Cancer (FACT-O)Version 1/23/07 - This is a relative quality of life assessment; 100 = Best, 0 = Worst. It was developed and validated with cancer patients and includes physical well being, social well being, emotional well being and relationship with doctor subscales and can be summed into one total quality of life score. It is a standardized scale which collects data (scores 1-4) from 47 questions. Answers are transformed into a number between 0-100. Mean was calculated by adding up the values of the scores and dividing by the number of scores.
Time Frame: Baseline, 3 Months Post Treatment, 6 Months Post Treatment
Measure: Mean (Full Range); unit: Scores on a Scale
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Scores on a Scale
  Baseline (rounded to nearest whole number) | 87 [53 to 108]
  3 Months (rounded to nearest whole number) | 84 [63 to 100]
  6 Months (rounded to nearest whole number) | 81 [79 to 96]

4. Secondary Outcome: Serum Skeletal-Specific Alkaline Phosphatase Concentration
Description: Median Bone mineral results - assessed by serum skeletal-specific alkaline phosphatase laboratory results collected from patients in study.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months
Measure: Median (Full Range); unit: Units/Liter
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Units/Liter
  Alkaline Phosphatase levels - Baseline | 14.0 [6.9 to 23.5]
  Alkaline Phosphatase levels - 1 Month | 16.1 [7.1 to 26.5]
  Alkaline Phosphase levels - 3 Months | 18.5 [8.3 to 25.5]
  Alkaline Phosphase levels - 6 Months | 16.2 [13.8 to 29.2]

5. Primary Outcome: Patients' Overall 90-Day Clinical Response as Measured by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Best response recorded from the start of treatment until Day 90. Defined by the sum of the Complete Responses (CR), Partial Responses (PR) and Stable Disease (SD) in patients treated with fulvestrant. CR=disappearance of all lesions, PR=>or =30% decrease in sum of all target lesions, Progressive Disease (PD) =>or=20% increase in sum of all target or any new lesions, SD=not CR, PR or PD.
Time Frame: Day 90
Measure: Number; unit: Participants
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Participants
  Stable Disease | 8
  Progressive Disease (>=20% increase/new lesions) | 18

6. Secondary Outcome: Urine N-telopeptide Concentration
Description: Median bone mineral results - assessed by serial urine N-telopeptide laboratory results collected from patients.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months
Measure: Median (Full Range); unit: Units of Bone Collagen Equivalents/mmol
Arm/Group | Fulvestrant Treatment
Number analyzed (Participants) | 26
Units of Bone Collagen Equivalents/mmol
  Urinary N-telopeptide level - Baseline | 50 [8 to 184]
  Urinary N-telopeptide level - 1 Month | 49 [11 to 117]
  Urinary N-telopeptide level - 3 Months | 43 [18 to 115]
  Urinary N-telopeptide level - 6 Months | 46 [42 to 91]

ADVERSE EVENTS:
Time Frame: Through 30 days after last treatment with Fulvestrant.
Arm/Group | Fulvestrant Treatment
Serious Adverse Events (participants affected / at risk) | 10/26
Other Adverse Events (participants affected / at risk) | 2/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Treatment (N=26)
Ascites (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bowel obstruction, non-specific (Gastrointestinal disorders) | 3 (3)
Death, non-specific (General disorders) | 2 (2)
Failure to thrive (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain, abdomen (General disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Treatment (N=26)
Bromidrosis (Skin and subcutaneous tissue disorders) | 2 (2) — Mild, foul smelling perspiration
Headache (Nervous system disorders) | 1 (1) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No